CLINICAL TRIAL: NCT04649411
Title: A 24-Week, Open-Label, Randomized, 2-Arm Study to Evaluate the Safety and Tolerability of KRX-0502 (Ferric Citrate) in Children With Iron Deficiency Anemia Associated With Non-Dialysis Dependent Chronic Kidney Disease
Brief Title: Study to Evaluate the Safety and Tolerability of KRX-0502 (Ferric Citrate) in Children With Iron Deficiency Anemia Associated With Non-Dialysis Dependent Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PMR release
Sponsor: Keryx Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRX-0502-309
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Iron Deficiency Anemia Associated With Non-Dialysis Dependent Chronic Kidney Disease
Keywords: Iron Deficiency Anemia; Non-Dialysis Dependent Chronic Kidney Disease; CKD; ferric citrate; pediatric; dialysis
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferric citrate; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ferric citrate (Experimental): Participants aged 12 to <18 years and 6 to <12 years will receive ferric citrate for 24 weeks at a starting dose based on body weight categories.
  Interventions: Drug: ferric citrate
- Standard of care (Active Comparator): Participants aged 12 to <18 years and 6 to <12 years will receive standard of care treatment for 24 weeks.
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: ferric citrate — oral tablets
  Other Names: KRX-0502
  Arms: Ferric citrate
Drug: standard of care — administered per the approved label and at the Investigator's discretion
  Arms: Standard of care

SUMMARY:
This study will be conducted to evaluate the safety and tolerability of ferric citrate in pediatric participants with iron deficiency anemia (IDA) associated with non-dialysis dependent chronic kidney disease (NDD-CKD).

ELIGIBILITY:
Inclusion Criteria:

* Age 6 years to <18 years at Screening
* Body Weight ≥12 kilograms (kg) at Screening
* Chronic kidney disease (CKD) stage 3 to 5, not on dialysis, with estimated glomerular filtration rate (eGFR) <60 milliliters per minute (mL/min)/1.73 meters squared (m^2) utilizing the "Bedside Schwartz" equation
* Hemoglobin (Hgb) ≥8.5 and ≤11.5 grams per deciliter (g/dL) at Screening
* Transferrin saturation (TSAT) ≤25% at Screening
* Ferritin ≤200 nanograms per milliliter (ng/mL) at Screening

Exclusion Criteria:

* Serum phosphorus level at Screening:

  * 6 to <13 years: ≤4.0 milligrams per deciliter (mg/dL);
  * 13 to <18 years: ≤2.7 mg/dL
* Liver transaminases (aspartate aminotransferase [AST] and/or alanine aminotransferase [ALT]) ˃3× the upper limit of normal at Screening
* Active significant gastrointestinal (GI) disorder, including overt gastrointestinal (GI) bleeding or active inflammatory bowel disease
* Unable to swallow pills
* Anemia due to causes other than iron deficiency anemia (IDA) of CKD
* Intravenous iron therapy or blood transfusion within 4 weeks before the Screening visit
* Participants with a functioning organ transplant
* Receipt of any investigational drug within 4 weeks before Screening
* Phosphate binder use during the Screening period

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Serious and Non-serious Treatment-emergent Adverse Events | up to Week 28
Number of Participants with Clinically Significant Laboratory Abnormalities or Changes in Laboratory Results | up to Week 24
Number of Participants with Treatment-emergent Adverse Events Leading to the Discontinuation of Ferric Citrate | up to Week 28

SECONDARY OUTCOMES:
Change from Baseline in Hemoglobin to Week 24/Early Termination Visit | Baseline; Week 24
Change from Baseline in Transferrin Saturation (TSAT) to Week 24/Early Termination Visit | Baseline; Week 24
Change from Baseline in Ferritin to Week 24/Early Termination Visit | Baseline; Week 24
Change from Baseline in Serum Phosphorus to Week 24/Early Termination Visit | Baseline; Week 24
Change from Baseline in Calcium to Week 24/Early Termination Visit | Baseline; Week 24
Change from Baseline in Bicarbonate to Week 24/Early Termination Visit | Baseline; Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.

IPD SHARING:
Plan to Share IPD: No